CLINICAL TRIAL: NCT02961569
Title: Comparative Study Between the Classical Strategy and a Faster, Daily Collection for the Diagnosis of Contagious Pulmonary Tuberculosis
Brief Title: Comparison Between Two Strategies for the Diagnosis of TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, Principal Investigator, Hopital Lariboisière
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TBsputum
Record Dates: First submitted 2016-10-18; First posted 2016-11-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary TB
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One open-label arm (Other): Patients suspected of pulmonary TB will have sputum collection for acid fast bacilli by the classical strategy (Day 1, Day 2 and Day 3) and the intervention sputum collection for acid fast bacilli by the same day strategy (Hour 1, 2 and 3)
  Interventions: Procedure: sputum collection for acid fast bacilli

INTERVENTIONS:
Procedure: sputum collection for acid fast bacilli — spontaneous or post fiberoptic bronchoscopy sputa

SUMMARY:
Tuberculosis (TB) is a major cause of death among the "communicable" diseases in the world. Pulmonary TB, the main localization, leads to the dissemination of cases. An earlier diagnosis of contagious pulmonary TB is a cornerstone to stop the air transmission. The aim of the study will be to compare two strategies, in patients with a chest-X-ray in favour of contagious pulmonary TB: the classical strategy of sputa collection during three consecutive early mornings, versus the studied strategy of sputa collection at hour h, hour h+1, hour h+2 during the first early morning.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major cause of death among the "communicable" diseases in the world. Pulmonary TB, the main localization, leads to the dissemination of cases. An earlier diagnosis of contagious pulmonary TB is a cornerstone to stop the air transmission by starting earlier treatment. The aim of the study will be to compare two strategies, in patients with a chest-X-ray in favour of pulmonary TB: the classical strategy of sputa collection during three consecutive early mornings, versus the studied strategy of sputa collection at hour h, hour h+1, hour h+2 during the first early morning.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients suspected of pulmonary TB (symptoms: lost weight, hemoptysis, chronic cough or fever, or a Chest-X-Ray (CXR) evocative of pulmonary TB)

Exclusion Criteria:

* Patients who refused or were unable to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Comparison between the sensitivities of the two strategies for detection of Acid fast bacilli (AFB) on direct stain | one year
  Ziehl Neelsen

CONTACTS AND LOCATIONS:
Overall Officials: Célia Lloret-Linares, MD, PhD, Principal Investigator — Unité de Recherches Thérapeutiques, Hôpital Lariboisière
Locations (1):
- Hôpital Lariboisière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes A, Mougari F, Chopin D, Pogliaghi M, Munier AL, Delcey V, Simoneau G, Raskine L, Evans J, Mouly S, Cambau E, Bergmann JF, Sellier P. Prospective study comparing the conventional and same-day strategies to diagnose pulmonary tuberculosis. Med Mal Infect. 2020 Feb;50(1):36-42. doi: 10.1016/j.medmal.2019.03.010. Epub 2019 Apr 11. PMID 30982671